CLINICAL TRIAL: NCT06780735
Title: Surgical Outcome of Breast Conserving Surgery Using Indocyanine Green Fluorescence in Breast Cancer Patients After Preoperative Chemotherapy: a Prospective Study
Brief Title: Surgical Outcome of BCS Using ICG-F in Breast Cancer Patients After Preoperative Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Seeyoun Lee, Doctor, M.D., head of center for breast cancer, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC-2310621-1
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Breast Neoplasms; Breast Cancer
Keywords: Indocyanine green; Breast conserving surgery; Breast cancer; neoadjuvant chemotherapy; Tumor Localization; Near-Infrared Fluorescence Imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ICG-F (Experimental): Localization of breast cancer using indocyanine green fluorescence (ICG-F)
  Interventions: Procedure: The margin-positive rate using the localization technique

INTERVENTIONS:
Procedure: The margin-positive rate using the localization technique — Localization of breast cancer using indocyanine green fluorescence (ICG-F)

SUMMARY:
Neoadjuvant chemotherapy for advanced breast cancer has led to an increased rate of breast-conserving surgery (BCS) in these patients. As the demand for preoperative localization methods grows among surgeons performing BCS, traditional localization techniques have shown limitations. For non-palpable breast lesions, preoperative localization has commonly been achieved using ultrasound-guided skin markings or needle localization. However, these methods present challenges, including difficulty in depth localization for patients with large breasts and limitations in real-time re-verification during surgery due to air artifacts after incision. Needle localization, although commonly used, is invasive and poses risks such as displacement or detachment of the needle.

Indocyanine green (ICG), a fluorescent dye that appears green to the naked eye and is detectable by near-infrared (NIR) cameras, has been widely and safely used in clinical practice via intravenous or subcutaneous administration. Recently, ICG combined with NIR imaging has been adopted for sentinel lymph node biopsy in breast cancer and melanoma surgeries and is increasingly used as a localization method for various tumors, replacing conventional techniques.

A preliminary study (IRB No. NCC2016-0071) conducted at the institution evaluated ICG injection and NIR fluorescence imaging for tumor localization in early breast cancer patients undergoing BCS. The study demonstrated the efficacy of ICG-based localization in reducing the rate of positive surgical margins.

The objective of this study is to evaluate the effectiveness of ICG-guided tumor localization with NIR fluorescence imaging in patients with advanced breast cancer treated with neoadjuvant chemotherapy. It is hypothesized that this technique will allow for more accurate tumor excision compared to conventional methods, ultimately improving surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* The Patient with locally advanced breast cancer who is eligible for breast-conserving surgery after receiving neoadjuvant chemotherapy
* Aged over 18 years old
* ECOG performance status: 0 or 1
* The patients with written informed consent

Exclusion Criteria:

* The patient who requires total mastectomy after receiving neoadjuvant chemotherapy
* The patient with no residual mass on ultrasonography or only with microcalcifications
* Pregnant or lactating patient
* The patient with a disability to understand and provide consent
* The patient with severe allergic history to indocyanine green
* Iodine-sensitive patient

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Margin-positive rate in final pathological report | 10~35 days after surgery (the date when the pathological reports are available)
  Collection of data for margin-positive rate from final pathological report after surgery

SECONDARY OUTCOMES:
Localization rate | The day of surgery
  Collection of data for tumor detection rate using ICG-F
Centralization | 10~35 days after surgery (the date when the pathological reports are available)
  Collection of data for the lengths from tumor to each resection margins
Margin-positive rate in frozen section | The day of surgery
  Collection of data for margin-positive rate in frozen section during surgery
Additional resection rate | The day of surgery
  Collection of data for additional resection rate according to results of frozen section during surgery
Re-excision rate | 10~35 days after surgery (the date when the pathological reports are available)
  Collection of data for re-excision rate (2nd operation) according to final pathological results
Adverse event rate | 10~35 days after surgery (the date of follow-up after surgery)
  Collection of data for pigmentation rate of the injection site

CONTACTS AND LOCATIONS:
Overall Officials: Seeyoun Lee, MD, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided